CLINICAL TRIAL: NCT06997978
Title: Efficacy of Tele-rehabilitation Intervention on Hand, Cognitive Functions & Depression of Hemiparetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Alshimy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Alshimy, Assistant professor of Physical Therapy, AlRyada University for Science & Technology
Organization: AlRyada University for Science & Technology (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004309
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hemiparesis
Keywords: Tele-rehabilitation; Hand functions; Cognitive functions; Depression; Hemiparesis
MeSH Terms: conditions — Paresis; Depression | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): study group A (n = 15) received the hand rehabilitation program through the Tele-rehabilitation program, a technological device. The rehabilitation was three times a week for a total of twelve weeks (36 sessions) following the conclusion of the rehabilitation program.
  Interventions: Other: Tele-rehabilitation; Other: Hand rehabilitation program
- Group B (Experimental): control group B (n = 15) received the same hand rehabilitation program at the physical therapy clinic. The rehabilitation was three times a week for a total of twelve weeks (36 sessions) following the conclusion of the rehabilitation program.
  Interventions: Other: Hand rehabilitation program

INTERVENTIONS:
Other: Tele-rehabilitation — Patients at the Telerehabilitation group are contacted via laptops that have cameras, microphones, and a reliable internet connection. The therapist's laptop camera is positioned so the patient may watch the therapist while the therapist demonstrates the exercises. After the therapist performs the exercise on himself, the patient must see the therapist via a laptop camera and then perform the same activity again.
  Arms: Group A
Other: Hand rehabilitation program — 1. Free exercises:
     1. Wrist flexion and extension 2. Wrist side movement 3. Thumb flexion and extension 4-Finger opposition 5. Palm up and down
  2. Ball exercises:
     1. Ball grip
     2. Finger flexion
     3. Thumb extend
     4. The pinch exercise
     5. Opposition 6- Side squeeze
     7. Extend out
  3. Household exercises
     1. Roll movement
     2. Wrist curl
     3. Extending the wrist
  4. Pen exercises
     1. Pinch and release
     2. Pen spine
  5. Exercises with coins
     1. Coin drop
     2. Coin stacking

SUMMARY:
Information and communication technologies (ICT) are used in telerehabilitation to deliver rehabilitation treatments to patients in their homes or other locations.

DETAILED DESCRIPTION:
Thirty hemiparetic patients with mild hand dysfunction of both sexes participated in the study (Age range was 45- to 55-year-old); 15 patients in the control group (GB) received a selected hand rehabilitation program, whereas 15 patients in the study group (GA) received telerehabilitation intervention. The 9HPT (Nine-hole peg test), FMUE (Fugl Meyer upper extremity), MOCA (Montreal cognitive assessment scale), REHACOM system, and the BECK DEPRESSION INVENTORY QUESTIONNAIRE were used to evaluate the patients in both groups before and after the treatment program began.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 45 and 55 were included in this study.
* Both men and women were among the patients. Patients with duration of illness between three to six months.
* According to the modified Ashworth scale (MAS), the patients' hand spasticity ranged from grade 1 to +1.
* The patients had a Fugl Myer upper extremity score of at least nine, indicating mild hand function. On the BECK DEPRESSION INVENTORY questionnaire, the patients' score ranged from 17 to 20 (Borderline clinical depression). Every patient had good vision and hearing.
* The patients successfully filled out the consent form and completed the assigned activities.
* In order to enable video communication while at home, patients need to have at least ten years of education to be able to use a smart device that is connected to the internet, such as a laptop, phone, or tablet.
* In addition to medical care, the patients shouldn't receive any other kind of treatment.
* The patients should be able to communicate and obey commands with ease. - - The patients' MMSE scores were over 21, indicating good cognitive abilities.

Exclusion Criteria:

* Individuals with unstable medical conditions, such as unstable angina, symptomatic heart failure, or uncontrolled diabetes mellitus or hypertension. - --- Patients who are unable to utilize the video communication device, have moderate to severe impairment of hand functions, or have any other pathology impacting hand function except stroke.
* Patients who have visual or hearing impairments.
* Patients who have communication issues or who have trouble understanding or obeying instructions.
* Individuals who have seizures or psychological disorders.
* Patients who have not had a stroke but have another illness that impairs cognitive function.
* Individuals who have a history of stroke or other neurological conditions.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
The Nine Hole Peg Test | 12 weeks
  Used to evaluate hemiparetic patients' finger dexterity
Fugl Myer Upper extremities | 12 weeks
  Intended to assess the motor functioning and impairment of stroke patients
Montreal Cognitive Assessment | 12 weeks
  Intended to identify moderate cognitive impairment and assess the various cognitive functions of stroke patients
REHACOM system | 12 weeks
  a software program made for diagnosing and treating patients with cognitive impairments. Figural memory (FM), attention concentration (AC), reaction behavior (RB), and logical reasoning (LR) are their four categories
Beck's Depression Inventory | 12 weeks
  a screening tool for depression and a means of determining the severity of depression

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ryada University for Science and Technology, Sadat, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No